CLINICAL TRIAL: NCT05907161
Title: The Effect of Low Laser Therapy and Hyaluronic Acid as an Adjunct to Non-surgical Periodontal Therapy in Patients With Periodontitis
Brief Title: Low Laser Therapy and Hyaluronic Acid as an Adjunct to Non-surgical Periodontal Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HA AND LASERS IN PERIO TH
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Before initial treatment the care provider will randomly pick an envelope with one of the three treatment modalities. At follow-up visits the investigator will perform the periodontal examination without having access to the patients data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- SRP (Experimental): The SRP group will receive non-surgical periodontal therapy using an ultrasonic device and curettes in two sessions.
  Interventions: Device: SRP
- SRP+LASER (Active Comparator): The SRP+LASER group will receive non-surgical periodontal therapy using an ultrasonic device and curettes in two sessions. After session 2, irradiation with a diode laser (Dentsply Sirona - SIROLaser Blue) will be applied intrasulcular to all sites with PD ≥ 4mm.
  Interventions: Device: SRP+LASER (Dentsply Sirona - SIROLaser Blue)
- SRP+HA (Active Comparator): The SRP+HA group will receive non-surgical periodontal therapy using an ultrasonic device and curettes in two sessions. After session 2, a gel containing hyaluronic acid (Regedent, HyaDENT Cross linked hyaluronic acid gel) will be applied intrasulcular to all sites with PD ≥ 4mm.
  Interventions: Device: SRP+HA

INTERVENTIONS:
Device: SRP+LASER (Dentsply Sirona - SIROLaser Blue) — adjunct irradiation with a diode laser (Dentsply Sirona - SIROLaser Blue) intrasulcularly to all sites with PD ≥ 4mm
  Arms: SRP+LASER
Device: SRP+HA — adjunct hyaluronic acid (Regedent, HyaDENT Cross linked hyaluronic intrasulcularly to all sites with PD ≥ 4mm
  Arms: SRP+HA
Device: SRP — non-surgical periodontal therapy (SRP) with utrasonic device and curretes
  Arms: SRP

SUMMARY:
Periodontal disease is an oral disease characterized by microbially associated, host-mediated inflammation of the periodontium. In the treatment of periodontal disease, conventional periodontal therapy includes both surgical and non-surgical approaches. Non-surgical therapy (i.e. scaling and root planing - SRP) remains an essential part of periodontal therapy. Here, diseased root surface debridement utilizing different hand and ultrasonic instrumentation is performed to facilitate periodontal re-attachment and to reduce the bacterial mass in the periodontal pocket.

In the last decade, the use of lasers (light amplification by stimulated emission of radiation) has occupied part of the dialogue within periodontology due to several proposed advantages. In the arena of periodontology, laser use, as an adjunct to non-surgical therapy, was demonstrated to enhance periodontal healing; however, it is still the matter of debate. Among laser applications, low-level laser therapy is recommended for its pain-reducing, woundhealing and anti-inflammatory effects.

Hyaluronic acid is a non-sulfated glycosaminoglycan and a major component of the extracellular matrix. It is found in various body fluids, such as gingival crevicular fluid, saliva, serum and synovial fluid. Anti-inflammatory, anti-edematous and anti-bacterial activities of hyaluronic acid have been investigated in dentistry, specially in periodontology.

DETAILED DESCRIPTION:
Each participant will be assigned in one of three groups. In each group there will be 15 participants. Different treatment protocols will be carried in each group as follows: group one (scaling and root planing), group two (scaling and root planing + LASER), group three (scaling and root planing + hyaluronic acid). Under local anesthesia we will perform scaling and root planing of the teeth in two sessions. The procedure be made with the use of ultrasonic (PiezoLED Scaler, KaVo, Biberach, DE) and hand instruments (Gracey, Hu Friedy, Chicago, IL, USA). In group one, only scaling and root planning (SRP) will be made. In group two, the use of a diode laser (Dentsply Sirona - SIROLaser Blue) will be added to the therapy. In group three, after the performance of SRP, a gel containing hyaluronic acid (Regedent, HyaDENT Cross linked hyaluronic acid gel) will be applied intrasulcular.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* nonsmokers
* untreated periodontal disease (stage 3, grade B or C)
* plaque index will not exceed 20%
* at least 20 teeth in oral cavity

Exclusion Criteria:

* systemic diseases with impact on periodontal health
* medication with impact on periodontal health
* smokers
* pregnant and lactating women
* patients treated with antibiotics in the last 12 months
* patients who had undergone periodontal treatment in the last year

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-06-09 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Probing pocket depth reduction | 3 months, 6 months
  Change in probing pocket depth after treatment

SECONDARY OUTCOMES:
Clinical attachment level gain | 3 months, 6 months
  Change in clinical attachment level after treatment
Bleeding on probing percentage reduction | 3 months, 6 months
  Bleeding after measurement of pocket depth, reduction after treatment
Residual diseased site number | 3 months, 6 months
  No of sites with PD ≥ 4mm and bleeding on probing after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Aleš Fidler, Dr., Study Director — University Medical Centre Ljubljana
Locations (1):
- Univerity Medical Center Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No